CLINICAL TRIAL: NCT02586194
Title: Pharmacokinetic Study of ASP015K - Evaluation of Pharmacokinetics in Patients With Impaired Hepatic Function and Subjects With Normal Hepatic Function
Brief Title: Pharmacokinetics Study in Patients With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 015K-CL-PK10
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2019-04

CONDITIONS: Patients With Impaired Hepatic Function
Keywords: Impaired hepatic function; Pharmacokinetics; ASP015K
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Subjects with normal hepatic function) (Experimental): Oral
  Interventions: Drug: ASP015K
- Mild hepatic impairment (Experimental): Oral
  Interventions: Drug: ASP015K
- Moderate hepatic impairment (Experimental): Oral
  Interventions: Drug: ASP015K

INTERVENTIONS:
Drug: ASP015K — Oral

SUMMARY:
The objective of this study is to compare and evaluate the pharmacokinetics of ASP015K in patients with impaired hepatic function and subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

A subject is eligible for the study if all of the following apply:

All subjects:

* Body weight: ≥40.0 kg and <90.0 kg
* Body mass index (BMI): ≥17.0 and <30.0 kg/m2
* Female subject must either:

  * Be post-menopausal or surgically sterile.
  * Agree not to try to become pregnant starting at the time of informed consent throughout the study period and for 60 days after the final study drug administration if she is of childbearing potential.
* Agrees to use highly effective contraception
* Agrees not to donate sperm (for male)/ ova (for female) starting at the time of informed consent, and throughout the study period and for 90/60 days after the final study drug administration.
* Female subject agrees not to breastfeed starting at the time of informed consent, and throughout the study period and for 60 days after the final study drug administration.
* Agrees not to participate in a clinical trial, a post-marketing study, or a clinical study during the period from informed consent to post examination.

A patient with impaired hepatic function:

* Impaired hepatic function Child-Pugh Score Class A (mild, 5-6 points) or Class B (moderate, 7-9 points).

A subject with normal hepatic function:

* Healthy, as judged by the investigator/subinvestigator based on physical examinations and all tests obtained at screening and during the period from hospital admission to immediately before study drug administration.

Exclusion Criteria:

A subject will be excluded from participation in this study if any of the following apply:

All subjects:

* Received or is scheduled to receive any investigational drugs in other clinical trials, post-marketing studies or clinical research within 120 days before screening or during the period from screening to the hospital admission.
* Excessive alcohol or smoking habit.
* Applies to any of following concerns of tuberculosis:

  * A history of active tuberculosis
  * Abnormalities detected on a chest X-ray test (at screening)
  * Contact with infectious tuberculous patients
* Applies to any of following concerns except for tuberculosis:

  * Concurrent or previous severe herpes zoster or herpes zoster disseminated
  * More than 1 recurrence of localized herpes zoster
  * Inpatient hospital care for severe infectious disease within 90 days before the hospital admission
  * Treatment with intravenous antibiotics within 90 days before the hospital admission (prophylactic antibiotics are not applicable)
  * Other than above, a people who has a risk of developing infectious diseases (e.g. urethral catheterisation) in judgment of the investigator/subinvestigator
* Vaccination of live vaccines or live attenuated vaccines within 56 days before the hospital admission (inactivated vaccines such as influenza vaccine and pneumococcal vaccine are not applicable).
* Concurrent or previous drug allergies.
* A history of clinically serious allergies (serious allergies: Generalised urticaria which requires hospital admission, allergy which causes anaphylactic shock, etc.).
* Concurrent or previous cardiac failure NYHA class 3 or 4, long QT syndrome and congenital short QT syndrome.
* Development of (an) upper gastrointestinal symptom(s) within 7 days before the hospital admission.
* Concurrent or previous lymphatic disease.
* A history of digestive tract excision, except for a history of appendectomy.
* Previous use of ASP015K.

A patient with impaired hepatic function:

* Unable to start washout of concomitant prohibited medications from at least 14 days prior to the study drug administration.
* Concurrent uncontrolled hypertension.
* Clinically significant abnormality detected on standard 12-lead electrocardiogram at screening or hospital admission.
* eGFR by the GFR estimating equation for Japanese <45 mL/min/1.73 m2 (the first decimal place rounded off) at screening.
* Uncontrolled ascites or pleural effusion observed at screening.
* Concurrent hepatic encephalopathy Coma Scale II or more at screening.
* Underwent hepatic transplantation, or underwent hepatectomy within 1 year before screening.
* Concurrent or previous drug-induced hepatic disorder.
* Concurrent acute hepatic disease.
* With surgically-placed portosystemic shunts including transjugular intrahepatic portosystemic shunts.
* Concurrent biliary obstruction.
* A history of oesophageal haemorrhage or gastric varices haemorrhage within 180 days before screening.
* Irregular or acute, and clinically significant LFT values or changes in clinical symptoms from 30 days before screening to immediately before study drug administration.
* Platelet count <4 × 104/μL, or haemoglobin <9 g/dL at screening.
* Alcohol dependence or unable to remain abstinent during the specified period.
* Concurrent esophagus or gastric varices which have a high risk of clinically significant haemorrhage.
* Concurrent cerebrovascular disorder, serious heart disease, malignant tumour or a history within 5 years before screening, gastrointestinal disease, urinary disease, renal disease, endocrine disease, and respiratory disease.

A subject with normal hepatic function:

* Received or is scheduled to receive medications (including over-the-counter drugs) within 7 days before the hospital admission.
* Deviates from any of the normal range of blood pressure, pulse rate, body temperature and standard 12-lead electrocardiogram at screening or the hospital admission.
* Meets any of the criteria for laboratory tests at screening or the hospital admission.
* eGFR by the GFR estimating equation for Japanese <60 mL/min/1.73 m2 (the first decimal place rounded off) at screening.
* Concurrent or previous hepatic disease, cerebrovascular disorder, malignant tumor, heart disease, gastrointestinal disease, except for a history of appendicitis, renal disease, endocrine disease, respiratory disease, urological disease.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of ASP015K: AUCinf | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72 hr after dosing
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameter of ASP015K: Cmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  Cmax: Maximum concentration
PK parameter of metabolites: AUCinf | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
PK parameter of metabolites: Cmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
Safety assessed by AEs | Up to 7 days after the study drug dosing
Safety assessed by Vital signs | Up to 7 days after the study drug dosing
  Supine blood pressure, supine pulse rate and axillary body temperature
Safety assessed by Laboratory tests | Up to 7 days after the study drug dosing
  Hematology, blood biochemistry, and urinalysis
Safety assessed by 12-lead ECGs | Up to 7 days after the study drug dosing

SECONDARY OUTCOMES:
PK parameters of ASP015K: AUClast | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  AUClast: Area under the concentration-time curve from the time of dosing extrapolated to the last measurable concentration
PK parameters of ASP015K: t1/2 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  t1/2: Terminal elimination half-life
PK parameters of ASP015K: tmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  tmax: Time of Cmax
PK parameters of ASP015K: CL/F | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  CL/F: Apparent total systemic clearance
PK parameters of ASP015K: Vz/F | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
  Vz/F: Apparent volume of distribution during the terminal elimination phase
PK parameters of metabolites: AUClast | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
PK parameters of metabolites: t1/2 | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing
PK parameters of metabolites: tmax | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 60 and 72hr after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Site JP00001, Fukuoka
  - Site JP00003, Kanagawa
  - Site JP00002, Tokyo
  - Site JP00004, Tokyo
  - Site JP00005, Tokyo
  - Site JP00006, Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Toyoshima J, Shibata M, Kaibara A, Kaneko Y, Izutsu H, Nishimura T. Population pharmacokinetic analysis of peficitinib in patients with rheumatoid arthritis. Br J Clin Pharmacol. 2021 Apr;87(4):2014-2022. doi: 10.1111/bcp.14605. Epub 2020 Dec 1. PMID 33068028